CLINICAL TRIAL: NCT04638738
Title: Implementation of Wearable Sensors and Digital Alerting Systems in Secondary Care: a Prospective Evaluation of Clinical Outcomes
Brief Title: Outcomes of Digital Alerting Systems in Secondary Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 17SM4043
Record Dates: First submitted 2020-11-10; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Sepsis; Deterioration, Clinical
Keywords: vital signs; continuous monitoring; wearable sensor
MeSH Terms: conditions — Sepsis; Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-implementation: Pre-implementation of digital alerting sensor systems
- Post-implementation: Implementation of digital alerting sensor systems
  Interventions: Device: SensiumVitals wearable patch sensor

INTERVENTIONS:
Device: SensiumVitals wearable patch sensor — Wearable sensor which measures heart rate, respiratory rate, and temperature continuously.
  Groups: Post-implementation

SUMMARY:
Why? The investigators are trying to find out if participants that suddenly deteriorate on the ward can be identified sooner by wearing a wearable sensor. This is an important study to see if the sensor works correctly in recording continuous vital observations of heart rate, respiratory rate and temperature. This information can help doctors and nurses identify un-well participants.

What? The investigators will ask the participants to wear a light wearable sensor on the chest that can be worn for 5 days. If the participants are still in hospital after this time the sensor can be changed. All sensors are disposable. The participants would not have to actively do anything to the sensor. We will also participants to complete a short questionnaire about the sensor.

Who? All participants on the ward that are admitted with a new medical or surgical problem can take part in the study. Participants undergoing a surgical procedure that require at least one overnight stay are eligible to take part in this study.

Where? This study is being conducted at West Middlesex University Hospital and St Marys Hospital Paddington. Only certain wards are being included at both sites, if the participant moves wards the sensor will be removed.

How? The study will last around 5 years and we aim to recruit 1000 participants.

ELIGIBILITY:
Inclusion Criteria:

* Admitted adults on a general medical or surgical ward, identified as suitable by the clinical team.
* Able to provide written consent

Exclusion Criteria:

* pacemaker/ICD
* open chest wound injury
* skin condition preventing sensor to be worn
* participant whom withdraws consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults admitted to general wards who will be staying at least 24h within hospital.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Time to acknowledge alert | through study completion, an average of 1 year
  Time to acknowledge alert on mobile device/central monitoring station

SECONDARY OUTCOMES:
Hospital length of stay | through study completion, an average of 1 year
  hospital length of stay
Mortality | through study completion, an average of 1 year
  Mortality within 30 days following discharge
Hospital readmissions | through study completion, an average of 1 year
intensive care step up | through study completion, an average of 1 year
  ITU step up

CONTACTS AND LOCATIONS:
Overall Officials: Meera Joshi, MRCS, PhD, Principal Investigator — Honorary research fellow
Locations (1):
- West Middlesex University Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iqbal FM, Joshi M, Fox R, Koutsoukou T, Sharma A, Wright M, Khan S, Ashrafian H, Darzi A. Outcomes of Vital Sign Monitoring of an Acute Surgical Cohort With Wearable Sensors and Digital Alerting Systems: A Pragmatically Designed Cohort Study and Propensity-Matched Analysis. Front Bioeng Biotechnol. 2022 Jun 27;10:895973. doi: 10.3389/fbioe.2022.895973. eCollection 2022. PMID 35832414
- [Derived] Joshi M, Ashrafian H, Arora S, Sharabiani M, McAndrew K, Khan SN, Cooke GS, Darzi A. A pilot study to investigate real-time digital alerting from wearable sensors in surgical patients. Pilot Feasibility Stud. 2022 Jul 6;8(1):140. doi: 10.1186/s40814-022-01084-2. PMID 35794669
- [Derived] Iqbal FM, Joshi M, Khan S, Ashrafian H, Darzi A. Implementation of Wearable Sensors and Digital Alerting Systems in Secondary Care: Protocol for a Real-World Prospective Study Evaluating Clinical Outcomes. JMIR Res Protoc. 2021 May 4;10(5):e26240. doi: 10.2196/26240. PMID 33944790